CLINICAL TRIAL: NCT05366569
Title: Bio-CAR-T Study on Pre and Post-infusion CAR-T Cell Therapy
Brief Title: Bio-CAR-T BS Study
Status: Recruiting | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Prof Domenico Russo, Head of Clinical Unit; Clinical Professor;, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: BIO-CAR-T BS 2022
Record Dates: First submitted 2022-04-22; First posted 2022-05-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL); Primary Mediastinal Large B-cell Lymphoma (PMBCL); Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection follow routinely timepoints for CAR-T Cell treatment monitoring. Therefore, the study is considered observational and not interventional.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this Study is the evaluation of post-infusion CAR-T (Chimeric Antigen Receptor T Cell) expansion and persistence in patients with DLBCL, PMBCL and ALL undergoing CAR-T therapy; and the feasibility and efficacy of the treatment in the real life practice.

DETAILED DESCRIPTION:
This Study is characterized by several biological sub-studies, reported as below:

* Post-infusion CAR-T expansion and persistence analysis by both Flow Cytometry and digital PCR (dPCR): the aim of this point are the evaluation and enumeration of CAR T cells (CD4+ and/or CD8+) during patients follow-up and set up of specific panels for longitudinal evaluation and monitoring of CAR-T subsets.
* Circulating Extracellular Vesicles quantification and analysis on peripheral blood and CNS (Central Nervous System) liquor: the aim are the identification of alterations in small EVs (Extracellular vesicles) ( number and cargos composition (proteins or miRNA) after CAR-T cell infusion and identification of small EVs markers which may distinguish patients "good responders" from patients "not responders" and/or which may predict particular post-infusion complications.
* Evaluation of neurological markers for ICANS (Immune effector cell-associated neurotoxicity syndrome): the purpose of this substudy are the assessment of previously identified plasma and CSF (Cerebrospinal fluid)biomarkers for inflammation, neuronal damage and glial activation in patients who develop ICANS and the characterize temporal neuronal and glial involvement by assessing plasma and CSF inflammatory, neuronal and glial biomarkers in ICANS and their role on outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-cell-ALL (≤ 25 years) or patients with DLBCL (18-70 years) or patients with PMBCL (18-70 years) who were relapsed/refractory after two lines of treatments;
* Adequate performance status (0 or 1);
* Adequate organ function;
* No active or uncontrolled infections;
* No thrombo-embolisms within the last 6 months;
* Absence of clinically relevant co-morbidities (e.g., select cardiovascular, neurologic, or immune disorders with organ dysfunction or requiring immunosuppressive treatment in the last 24 months);
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Patients with B-cell-ALL > 25 years
* Patients with DLBCL <18 or >70 years
* Patients with PMBCL <18 or >70 years
* Performance status > 1;
* Active or uncontrolled infections;
* Thrombo-embolisms within the last 6 months;
* Presence of clinically relevant co-morbidities (e.g., select cardiovascular, neurologic, or immune disorders with organ dysfunction or requiring immunosuppressive treatment in the last 24 months);
* Life expectancy < 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Calculation is based on the primary endpoints, i.e. the persistence of the CAR-T cells and the percentage of patients infused. As the Investigator have no formal statistical hypothesis to test, sample size justification is based on estimating the 95% confidence interval for the above percentage. Based on the UOC Hematology and Pediatric Oncohematology's experience and accrual potential, the Investigators are expecting about 180 patients newly diagnosed with DLBCL or PMBCL or ALL (potential candidate to CAR-T therapy) in a 3-year time window. About 25% of these patients are expected to be eligible to CAR T-cell treatment, corresponding to 45 patients. Thus, assuming a 25% percentage of patients infused, a sample size of 45 patients will produce a two-sided 95% confidence interval ranging from 12% to 38%, with a precision (half-width of 95% confidence interval) equal to 13%.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of change post-infusion CAR-T cell expansion and persistence in patients with DLBCL, PMBCL and ALL undergoing CAR-T therapy evaluated by flow-cytometry and measures by number of cells/mL | At day +1; +3; +7; +10; +14; +21; +30; +60; +90; +120; +150; +180; +210; +240; +270; +300; +330; +360 post CAR-T cell infusion or at any time for relapse/CRS-ICANS onset (assessed up to 2 years))
Change of disease burden after CAR-T Cells treatment | At day +30; +90; +180; 270 and + 360 post CAR-T infusion
  Disease response will be evaluated according to Lugano criteria

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v 4.0 and ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells | At day +1; +3; +7; +10; +14; +21; +30; +60; +90; +120; +150; +180; +210; +240; +270; +300; +330; +360 post CAR-T cell infusion or at any time for relapse/CRS-ICANS onset (assessed up to 2 years)
  CTCAE v 4.0 and ASTCT (American Society for Transplantation and Cellular Therapy) Consensus Grading for Cytokine Release Syndrome (CRS) and Neurologic Toxicity Associated with Immune Effector Cells
Evaluation of disease persistence and immune recovery and neurological biomarkers after CAR-T infusion | Before starting the treatment and at day +1; +3; +7; and +30 after infusion of CAR-T cell and in case of development of neurological symptoms
  In addiction to cytokine panel (IL-1, IL-2, IL-5, IL-6, IL-7, IL-10, IL-12, IL-15, IL-17A, GM-CSF, TNFα, IFNγ, IL-22, IL-23) as per normal clinical practice the investigators will process interleukin: IL 8, IL 1β and CP-1.
  Cytokine profiles will be analyzed from blood and CSF samples using Luminex platform and all the measure element will expressed in pg/mL.
Evaluation of plasma level of biomarkers for ICANS neural damage and glial activation in patients who develop ICANS. | Before starting the treatment and at day +1; +3; +7; and +30 after infusion of CAR-T cell and in case of development of neurological symptoms
  Evaluation of previously identify plasma and CSF biomarkers for inflammation,neural damage and glial activation in patients who develop ICANS.
  NfL and GFAP markers of neuronal injury and astroglia will be analyzed by SIMOAQuanterix, while sTREM2 (microglia activation) by Luminex, together with cytokines analysis.
  The unit of measurement will be pg/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, Italy

REFERENCES:
- [Derived] Farina M, Chiarini M, Almici C, Accorsi Buttini E, Zuccala F, Piva S, Volonghi I, Poli L, Bernardi S, Colnaghi F, Re F, Leoni A, Polverelli N, Turra A, Morello E, Galvagni A, Moratto D, Brugnoni D, Cattaneo C, Ferrari E, Bianchetti A, Malagola M, Re A, Russo D. Timely Leukapheresis May Interfere with the "Fitness" of Lymphocytes Collected for CAR-T Treatment in High Risk DLBCL Patients. Cancers (Basel). 2022 Oct 27;14(21):5276. doi: 10.3390/cancers14215276. PMID 36358694